CLINICAL TRIAL: NCT06048692
Title: The Impact of Cefepime and Unictam on Preventing Post-Cesarean Surgical Site Infections
Brief Title: Cefepime and Unictam on Preventing Post-Cesarean Surgical Site Infections
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: maxipime in cs
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Section; Infection
Keywords: surgical site infection; Cefepime
MeSH Terms: conditions — Infections; Surgical Wound Infection | interventions — Cefepime; sultamicillin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefepime Group (Experimental): Pregnant women (n=100) received IV cefepime (CEF) (maxipime®1000mg) 30 minutes before cesarean delivery (CD) and 12 hours after CD
  Interventions: Drug: Cefepime 1000 MG
- Ampicillin/Sulbactam (Active Comparator): Pregnant women (n=100) received IV Ampicillin/Sulbactam (AMS) (Unictam® 1500 mg) 30 minutes before CD and 12 hours after CD
  Interventions: Drug: Ampicillin-sulbactam

INTERVENTIONS:
Drug: Cefepime 1000 MG — Cefepime is a fourth-generation cephalosporin antibiotic
  Other Names: maxipime
  Arms: Cefepime Group
Drug: Ampicillin-sulbactam — Broad-Spectrum Antibiotic
  Other Names: unictam
  Arms: Ampicillin/Sulbactam

SUMMARY:
the aim of this study is to evaluate the efficacy of employing cefepime (CFM) versus ampicillin/sulbactam (AMS) in lowering the rate of post-cesarean surgical site infections.

DETAILED DESCRIPTION:
A prospective randomized clinical study conducted in the department of obstetrics and gynecology of Beni-Suef University Hospital . A total of 213 women were assessed for eligibility, 13 of which were excluded. A total of 200 pregnant women who were eligible for elective cesarean sections (CS). The overall median duration of postoperative followed up was from 10 days to one month to determine the surgical site infection (SSI).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women within age group more than18 years.
* Pregnant women with elective cesarean delivery.
* Previous and primary cesarean delivery.

Exclusion Criteria:

Severe hepatic disease women Emergent cesarean deliveries. Women with medical disorders as pre-gestational diabetes, anemia, hypertension, or preeclampsia.

Women who had a skin infection adjacent to the operative site.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
surgical site infection | 1 month
  pain, redness, swelling, warm skin around the wound, yellow or green discharge

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided